CLINICAL TRIAL: NCT03454529
Title: The Effect of Statins on Markers of Breast Cancer Proliferation and Apoptosis in Women With Early Stage Breast Cancer
Brief Title: The Effect of Simvastatin on Breast Cancer Cell Growth in Women With Stage I-II Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Michael Simon (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Michael Simon, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Organization: Barbara Ann Karmanos Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-073; NCI-2018-00044 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-073 (Other: Wayne State University/Karmanos Cancer Institute); P30CA022453 (NIH)
Record Dates: First submitted 2018-02-22; First posted 2018-03-06 (Actual); Results first posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Invasive Breast Carcinoma; Stage I Breast Cancer AJCC v7; Stage IA Breast Cancer AJCC v7; Stage IB Breast Cancer AJCC v7; Stage II Breast Cancer AJCC v6 and v7; Stage IIA Breast Cancer AJCC v6 and v7; Stage IIB Breast Cancer AJCC v6 and v7
MeSH Terms: conditions — Breast Neoplasms | interventions — Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (simvastatin) (Experimental): Patients receive simvastatin PO daily for 2-4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Simvastatin

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Simvastatin — Given PO
  Other Names: MK 733; Synvinolin; Zocor

SUMMARY:
The purpose of this pilot phase II trial is to identify the molecular and genetic mechanisms by which statins influence breast cancer cell proliferation. Simvastatin may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and reduce the aggressiveness of breast cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the relationship between short-term use of oral simvastatin on change in expression of Ki-67 as a candidate biomarker of breast tumor proliferation among women with clinical stage 1 or 2- primary invasive breast cancer.

II. Evaluate the relationship between short-term use of oral simvastatin on changes in other candidate predictive markers of breast tumor proliferation (cyclin D1 and P27), changes in a marker of apoptosis (cleaved caspase-3 [CC3]), changes in a marker of inflammation (c-reactive protein [CRP]) and as novel additional biomarkers changes in the composition of the plasma membrane (lipid rafts) and changes in activation of signaling markers (phosphorylation [p]Akt, pMAPK, pEGFR, PHER2).

III. To conduct exploratory analyses comparing the effect of statins on breast tumor proliferation and apoptosis in groups defined by tumor expression of hydroxymethylglutaryl co-enzyme A (CoA) reductase (HMG-CoA), estrogen receptor (ER)/progesterone receptor (PR) status, HER2neu, and tumor grade.

OUTLINE:

Patients receive simvastatin orally (PO) daily for 2-4 weeks in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Histologic confirmation of invasive breast cancer with any measures of ER, PR and HER2neu
* Clinical stage I or II breast cancer for which there will be at least a 2 week period of time between diagnosis and definitive surgery
* Performance status (Eastern Cooperative Oncology Group [ECOG] 0-1)
* Not currently pregnant during the study; participants will be informed that the use of contraceptive pills is contraindicated because it may interfere with the study drug and it may be harmful to the woman who has been diagnosed with breast cancer

Exclusion Criteria:

* Plans for administration of neoadjuvant chemotherapy or hormonal therapy
* Insufficient tissue on diagnostic core breast biopsy for analysis
* Previous or concurrent malignancy (with the exception of non-melanomatous skin cancer)
* Severe gastrointestinal disorder
* Current use of statins or fibrates for any time during the 3 months prior to the study
* Proven hypersensitivity to statins
* White blood cell (WBC) < 3,500/mm^3
* Platelet (Plt) < 120,000/mm^3
* Hemoglobin (HgB) < 10 g/dL
* Aspartate aminotransferase (AST) > 45 U/L
* Alanine aminotransferase (ALT) > 45 U/L
* Creatinine > 1.5 mg/dL
* Bilirubin > 1.15 mg/dL
* Creatine kinase measurement (CPK) > or = 250 mg/dL
* Central nervous system (CNS) diseases and major psychiatric diseases or inability to comply to the protocol procedures
* Active infections
* Cardiac failure, class I-IV
* Current anticoagulant or antiplatelet aggregation therapy
* Mitral and/or tricuspid valvopathy or valvular prosthesis; angina; severe arterial hypertension; chronic and/or paroxysmal atrial fibrillation; previous myocardial infarction
* Current lactation

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-03-09 (Actual); Primary Completion 2021-10-06 (Actual); Study Completion 2021-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Simon, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Wayne State University/Karmanos Cancer Institute, Detroit, Michigan, United States

REFERENCES:
- [Derived] Asari K, Sun WT, Kok ZH, Lam YH, Ng BL, Saunders V, White DL, Chuah C, Xiang W. Simvastatin enhances the efficacy of nilotinib in chronic myeloid leukaemia by post-translational modification and drug transporter modulation. Anticancer Drugs. 2021 Jun 1;32(5):526-536. doi: 10.1097/CAD.0000000000001028. PMID 33587350

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Simvastatin)
Started | 24
Completed | 17
Not Completed | 7
Not completed — Did not receive treatment | 6
Not completed — Received < 80% doses | 1

BASELINE CHARACTERISTICS:
Population: All evaluable patients, including those recevied >80% doses
Arm/Group | Treatment (Simvastatin)
Number analyzed (Participants) | 17
Age, Continuous [Median (Full Range); unit: years] | 63 [48 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 9
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  United States | 17
Estrogen Receptor Status [Count of Participants; unit: Participants]
  Positive | 15
  Negative | 2
Progesterone Receptor Status [Count of Participants; unit: Participants]
  Positive | 11
  Negative | 6
HER2 Status [Count of Participants; unit: Participants]
  Positive | 0
  Negative | 12
  Unknown | 5
Tumor Stage [Count of Participants; unit: Participants] — Stage 0: In Situ; the cancer is limited to the inside of the milk duct and is non-invasive (does not invade nearby tissues).
  Stage I: Invasive; Primary Tumor < 20mm; No lymph nodes affected; No metastasis Stage II: Invasive: Primary Tumor 20-50 mm; No lymph node involvement OR lymph node involvement of < 4 lymph nodes in the same side of the breast; No metastasis
  Participants
    Stage 0: limited to the inside of the milk duct; is non-invasive; does not invade nearby tissues. | 6
    Stage I: Invasive; Primary Tumor < 20mm; No lymph nodes affected; No metastasis. | 11
    Stage II: Primary Tumor 20-50 mm; 0-<4 lymph nodes in the same side of the breast; No metastasis | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Ki-67 Expression Assessed in Tumor Tissue by Immunohistochemistry
Description: Differences in % positive cells pre and post treatment along with 95% confidence interval
Time Frame: Baseline up to 4 weeks
Population: one patient did not have pre and post measures
Measure: Mean (95% Confidence Interval); unit: percentage of cells expressing Ki67
Arm/Group | Treatment (Simvastatin)
Number analyzed (Participants) | 16
percentage of cells expressing Ki67 | 1.3 [-3.6 to 6.2]

2. Other Pre Specified Outcome: Change in Percentage of Cells P27+ From Pre-treatment to Post-treatment
Description: The difference in percentage of cells P27+ from pre-treatment to post-treatment
Time Frame: Baseline up to 4 weeks
Measure: Mean (95% Confidence Interval); unit: percentage of cells 'biomarker' positive
Arm/Group | Treatment (Simvastatin)
Number analyzed (Participants) | 16
percentage of cells 'biomarker' positive | -1.4 [-9.2 to 6.3]

3. Other Pre Specified Outcome: Cleaved Caspase-3 (CC3) as a Marker of Apoptosis
Description: The difference in (percentage of cells cleaved caspase-3 (CC3)+) from pre-treatment to post-treatment
Time Frame: Baseline up to 4 weeks
Measure: Mean (95% Confidence Interval); unit: percentage of cells expressing CC3
Arm/Group | Treatment (Simvastatin)
Number analyzed (Participants) | 16
percentage of cells expressing CC3 | 5.4 [-1.3 to 12.1]

4. Other Pre Specified Outcome: C-reactive Protein (CRP) as a Marker of Inflammation
Description: c-reactive protein (CRP) as a marker of inflammation.
Time Frame: Baseline up to 4 weeks
Population: This biomarker was not measured.
Arm/Group | Treatment (Simvastatin)
Number analyzed (Participants) | 0

5. Other Pre Specified Outcome: Change in (% Intracellular p27 +) From Pre-treatment to Post-treatment
Description: the difference in (% intracellular p27 +) from pre-treatment to post-treatment
Time Frame: Baseline up to 4 weeks
Measure: Mean (95% Confidence Interval); unit: percentage of intracellular p27 +
Arm/Group | Treatment (Simvastatin)
Number analyzed (Participants) | 16
percentage of intracellular p27 + | 0.3 [-7.9 to 8.4]

6. Other Pre Specified Outcome: Changes in p27 Cytoplasmic Intensity
Description: the difference in (p27 cytoplasmic intensity) from pre-treatment to post-treatment
Time Frame: Baseline up to 4 weeks
Measure: Mean (95% Confidence Interval); unit: arbitrary units
Arm/Group | Treatment (Simvastatin)
Number analyzed (Participants) | 16
arbitrary units | 1.8 [0.2 to 3.4]

7. Other Pre Specified Outcome: Changes in Cyclin D1
Description: the difference in % cyclin D1+ stained out of total cells from pre-treatment to post-treatment;
Time Frame: Baseline up to 4 weeks
Population: all 16 evaluable participants, except that one patient's sample did not yield cyclin D1 measurement.
Measure: Mean (95% Confidence Interval); unit: percentage of total cells cyclin +
Arm/Group | Treatment (Simvastatin)
Number analyzed (Participants) | 15
percentage of total cells cyclin + | 6.1 [-2.1 to 14.2]

ADVERSE EVENTS:
Time Frame: from enrollment up to 18 months
Arm/Group | Treatment (Simvastatin)
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 2/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Simvastatin) (N=17)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/29/NCT03454529/Prot_SAP_001.pdf